CLINICAL TRIAL: NCT00177476
Title: Enhancing Exercise Participation in Overweight Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HL067826-01A2 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

INTERVENTIONS:
Behavioral: behavioral weight loss

SUMMARY:
The purpose of this study is to examine whether behavioral strategies implemented during the adoption versus the maintenance periods of weight loss to enhance exercise participation in overweight adults are more effective than a standard behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male
2. 18-55 years of age
3. BMI = 25-39.9 kg/m2
4. Ability to provide informed consent.
5. Ability to provide consent from their personal physician to participate in this study.

Exclusion Criteria:

1. Reporting regular exercise participation of at least 20 minutes per day on at least 3 days per week during the previous six months. (This study is designed to recruit relatively sedentary adults.)
2. Diabetes, hypothyroidism, or other medical conditions which would affect energy metabolism.
3. Women who are currently pregnant, pregnant within the previous six months, or planning on becoming pregnant within the next 18 months. (Pregnancy during initial screening will be based on self-report and will be included on the detailed medical history that is completed by subjects)
4. Non-medicated resting systolic blood pressure >160 mmHg or non-medicated resting diastolic blood pressure >100 mmHg, or taking medication that would affect blood pressure.
5. Taking medication that would affect resting heart rate or the heart rate response during exercise (e.g., beta blockade).
6. Arrhythmia on resting or exercise electrocardiogram that would indicate that vigorous exercise was contraindicated.
7. History of myocardial infarction or valvular disease.
8. Weight loss of >5% of body weight within the previous 12 months.
9. History of orthopedic complications that would prevent optimal participation in the exercise component (e.g., heel spurs, severe arthritis).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225
Dates: Start 2003-09; Study Completion 2006-05

PRIMARY OUTCOMES:
body weight

SECONDARY OUTCOMES:
Fitness
physical activity
dietary intake
mediators

CONTACTS AND LOCATIONS:
Overall Officials: John M. Jakicic, Ph.D., Principal Investigator — University of Pittsburgh

REFERENCES:
- [Derived] Jakicic JM, Rickman AD, Lang W, Davis KK, Gibbs BB, Neiberg R, Marcus MD. Time-based physical activity interventions for weight loss: a randomized trial. Med Sci Sports Exerc. 2015 May;47(5):1061-9. doi: 10.1249/MSS.0000000000000482. PMID 25160843
- [Derived] Janney CA, Jakicic JM. The influence of exercise and BMI on injuries and illnesses in overweight and obese individuals: a randomized control trial. Int J Behav Nutr Phys Act. 2010 Jan 6;7:1. doi: 10.1186/1479-5868-7-1. PMID 20145731